CLINICAL TRIAL: NCT06860893
Title: Spinal Anesthesia as an Adjunct to General Anesthesia for Robotic Assisted Laparoscopic Prostatectomy - a Randomised Placebo- Controlled Trial
Brief Title: Spinal Anesthesia for Robotic Assisted Laparoscopic Prostatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Prostate REK 866656
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer Surgery
Keywords: Spinal anesthesia; Robotic assisted prostatectomy; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Double blinded placebo controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal anesthesia (Active Comparator): After obtaining return of cerebrospinal fluid, hyperbaric bupivacaine 5 mg/mL 1,5 mL (7,5 mg) and morphine 200 µg/mL, 0.5 mL (100 µg) was injected intrathecally.
  Interventions: Drug: Spinal Anesthesia with Bupivacaine
- Placebo (Placebo Comparator): Local skin infiltration with lidocain 10 mg/ml
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spinal Anesthesia with Bupivacaine — After obtaining return of cerebrospinal fluid, hyperbaric bupivacaine 5 mg/mL 1,5 mL (7,5 mg) and morphine 200 µg/mL, 0.5 mL (100 µg) was injected intrathecally.
  Arms: Spinal anesthesia
Drug: Placebo — Local skin infiltration with lidocaine
  Arms: Placebo

SUMMARY:
The investigators hypothesised that spinal anesthesia as an adjunct to general anesthesia would facilitate faster recovery and less pain in patients undergoing laparoscopic robotic prostatectomy. A double-blind placebo-controlled study was subsequently designed.

DETAILED DESCRIPTION:
Patients were allocated to either intrathecal injection of bupivacaine/morphine or a sham spinal procedure. All patients were placed in a sitting position and the skin over the lumbar region of the back was disinfected with chlorhexidine and draped sterile. In the intervention group the skin was infiltrated with 5 mL of lidocaine 10 mg/mL and a sterile 27-gauge pencil-point needle (Pajunk, GA, USA) was subsequently entered into the intrathecal space at the L2-3 or L3-4 interspace. After obtaining return of cerebrospinal fluid, hyperbaric bupivacaine 5 mg/mL 1,5 mL (7,5 mg) and morphine 200 µg/mL, 0.5 mL (100 µg) was injected intrathecally. Patients in the placebo group received an identical treatment as the patients in the intervention group, except for the intrathecal injection. After the skin was infiltrated with 5 mL of lidocaine 10 mg/mL, the attending anesthesiologist pressed one finger at the skin and talked as if she was giving an intrathecal injection at the L3-4 interspace. All patients were treated by the same anesthesiologist (MA).

ELIGIBILITY:
Inclusion Criteria:

- Prostate cancer

Exclusion Criteria:

* Benign prostate disease

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 30 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Time to discharge from the post anesthesia care unit. | 24 hrs
  Minutes of stay in the post anesthesia care unit

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of North Norway, Tromsø, Norway